CLINICAL TRIAL: NCT05329519
Title: The Effects of Listening Music During Breathing Exercises on Vital Sings and Pulmonary Functions After Video-assisted Thoracoscopic Surgery:A Randomized-controlled Study
Brief Title: The Effects of Listening Music During Breathing Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Collaborators: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Ozgu Bakcek, Lecturer, RN, MSc, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YuksekIhtisas
Record Dates: First submitted 2022-03-22; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Perioperative Complication; Nursing Caries; Pain, Postoperative
Keywords: Nursing; Thoracic surgery; Listening music; Deep breathing and coughing exercise; Pulmonary function; Vital signs
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: 2 parallel group randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): Patients in this groups underwent VATS with wedge recession, performed deep breathing and coughing exercises while listening to music for thirty minutes a day with a MP3 player and head phones on postoperative three days.
  Interventions: Behavioral: Listening music
- Controlled group (No Intervention): Patients in this groups underwent VATS with wedge recession, performed deep breathing and coughing exercises for postoperative three days without music

INTERVENTIONS:
Behavioral: Listening music — Patients in both groups underwent VATS with wedge recession and the same surgical methods were employed. After the surgery, the patients in the music group performed deep breathing and coughing exercises while listening to music for thirty minutes a day with a MP3 player (Goldmaster Goldsmart Mp3-159 Player) and head phones on postoperative days 1, 2, and 3. We prepared a list of popular songs of different genres, including Turkish classical, folk, pop and rock music, classical music and foreign music, and allowed them to choose the song to be listened.
  Other Names: Music group
  Arms: Music group

SUMMARY:
Background and purpose : This study aims to analyze the effects of listening to music during deep breathing and coughing exercises on vital sings and pulmonary functions in patients, who underwent video assisted thoracoscopic surgery with wedge resection.

Materials and methods: This randomized and single-blinded study was conducted on 30 patients, including 15 patients in the music and the control groups. The patients were randomized into the music group, which listened to music during deep breathing and coughing exercises and the control group that only performed the exercises. Data were collected preoperatively and postoperatively. Patient information form, observation form and the visual analog scale were used for data collection.

DETAILED DESCRIPTION:
2. Methods 2.1. Study design and setting This randomized trial was conducted at a research and training hospital in Ankara province of Turkey between June 2016 and January 2017.

2.2. Sample size Sample size was calculated with reference to the change in pain scores in a study of (music group: 29.7 ± 19.8, control group: 50.7±19.2). A total of 22 patients with 11 in each group were needed for Type I error of 0.05 and Type II error of 0.20. Given the possibility of withdrawals, study was intended to reach 30 patients with 15 in each group.

Since the patients in the control and intervention (music) groups could share their experiences before the surgery, randomized the patients weekly. With this aim, 'R Studio' software was used for block randomization to determine the groups that would receive the intervention on each week. The patients were single-blinded so that they were unaware of which group they had been assigned to.

Study included the voluntary patients age of 18 years and above the age of 18 years, who would undergo a video assisted thoracoscopic surgery with wedge resection, could read and write in Turkish, had no visual and auditory problems, and were categorized as ASA I, ASA II or ASA III patients according to the American Society of Anesthesiologists (ASA) physical status classification system. Patients with visual and auditory problems, who could not read or write in Turkish and priorly underwent a video assisted thoracoscopic surgery with wedge resection were excluded.

2.3. Tools Patient information form, observation from and the visual analog scale were used for data collection, which took place before the surgery and days 1, 2 and 3 postoperatively.

2.3.1. Patient Information Form The patient form was prepared by the researchers in line with the literature included four questions on the sociodemographic characteristics, such as age, gender, education level and working status, and two questions on the clinical characteristics, including, smoking and previous surgeries.

2.3.2. Observation Form The observation form was prepared by the researchers based on the literature and was used to record vital signs, such as. systolic and diastolic blood pressure (BP), heart rate, and the parameters of pulmonary functions, including forced vital capacity (FVC), forced expiratory volume in one second (FEV1) and the ratio of FEV1 to FVC (FEV1/FVC).

2.3.3. Visual Analog Scale (VAS) The VAS, which is frequently used in clinical practice to evaluate pain, was first developed in 1992. VAS is usually a 10 cm (100mm) long horizontal or vertical line and the responses range from 'no pain' to 'worst pain'. It may be a straight line or may be divided into equal intervals. Patients put a cross on at the point that most accurately expresses their degree of pain. The validity and reliability of the Turkish version was confirmed in 2004.

2.4. Interventions Data were collected before and after the surgery. During the face-to-face interviews before the surgery, patients were informed about the aim of the study, gathered information on their sociodemographic and clinical characteristics, recorded vital signs and parameters about pulmonary functions and asked the patients to complete the VAS. Next, Patients were explained the importance of deep breathing and coughing exercises and demonstrated how to perform these exercises. Finally, delivered a booklet on the exercises, which was prepared by the researchers based on the literature.

Patients in both groups underwent video assisted thoracoscopic surgery with wedge recession and the same surgical methods were employed. After the surgery, the patients in the music group performed deep breathing and coughing exercises while listening to music for thirty minutes a day with a MPEG player 3 (Goldsmart Mp3-159 Player) and head phones on postoperative days 1, 2, and 3. A list of popular songs of different genres, including Turkish classical, folk, pop and rock music, classical music and foreign music, prepared and allowed them to choose the song to be listened. The patients in the controlled group, on the other hand, performed deep breathing and coughing exercises for three days without music. Vital signs and the parameters of pulmonary functions were recorded after each exercise.

The impact of music during deep berating and coughing exercises on vital signs and the parameters of pulmonary functions were recorded on postoperative days 1, 2 and 3. Datex Ohmeda (GE Healthcare, Finland) was used to measure vital signs, including heart rate, oxygen saturation and systolic and diastolic BP. Parameters of pulmonary functions were measured using One-Flow FVC Kit (3141001USB), and spirometer (Clement Clark Int.). A VAS was used to evaluate the intensity of pain.

2.5. Statistical analysis Statistical Package of Social Sciences (SPSS, Inc., Chicago, USA) version 15.0 was used for the analysis of collected data. As descriptive statistics, number (n) and frequency (%) were used for categorical variables while mean median and standard deviation were calculated for continuous variables. Shapiro-Wilk test was used to test the normality of the data. For intergroup comparison, we used the independent sample t-test if the data met normal distribution and the Mann-Whitney U-Test if the data did not meet normal distribution. The chi-square and Fisher's exact test were used to test for differences between categorical variables. Statistical significance was set at p < 0.05.

2.6. Ethical Considerations Before conducting this study, received permission from the ethical committee of the university (No. 50687469-1491-15-16/1648.4-115). The trial was conducted in accordance with the principles of Helsinki Declaration and verbal and written informed consent from all patients was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary patients
* Age of 18 years and above the age of 18 years, who would undergo a video assisted thoracoscopic surgery with wedge resection,
* Patient could read and write in Turkish,
* Patient had no visual and auditory problems,
* Patient were categorized as ASA I, ASA II or ASA III patients according to the American Society of Anesthesiologists (ASA) physical status classification system.

Exclusion Criteria:

* Non-voluntary patients
* Under the age of 18 years
* Patients with visual and auditory problems, who could not read or write in Turkish
* Patients priorly underwent a VATS with wedge resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | through study completion, an average of 6 months
  mm Hg (millimeters of mercury)
diastolic blood pressure | through study completion, an average of 6 months
  mm Hg (millimeters of mercury)

SECONDARY OUTCOMES:
forced vital capacity (FVC) | through study completion, an average of 6 months
  Liter/Second
forced expiratory volume in one second (FEV1) | through study completion, an average of 6 months
  Liter/Second

CONTACTS AND LOCATIONS:
Overall Officials: Sevinc Tastan, Proffessor, Study Director — Eastern Mediterrean University
Locations (1):
- Özgü Bakçek, Ankara, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campos JH, Peacher D. Choosing the Best Method for Postoperative Regional Analgesia After Video-Assisted Thoracoscopic Surgery. J Cardiothorac Vasc Anesth. 2020 Jul;34(7):1877-1880. doi: 10.1053/j.jvca.2020.02.043. Epub 2020 Feb 29. No abstract available. PMID 32253088
- [Background] Agostini PJ, Lugg ST, Adams K, Smith T, Kalkat MS, Rajesh PB, Steyn RS, Naidu B, Rushton A, Bishay E. Risk factors and short-term outcomes of postoperative pulmonary complications after VATS lobectomy. J Cardiothorac Surg. 2018 Apr 12;13(1):28. doi: 10.1186/s13019-018-0717-6. PMID 29673386
- [Background] Federici S, Gonzalez M. Uniportal video-assisted thoracoscopic right upper sleeve lobectomy. Multimed Man Cardiothorac Surg. 2019 Nov 26;2019. doi: 10.1510/mmcts.2019.043. PMID 31990152
- [Background] Gupta S, Groen RS, Kyamanywa P, Ameh EA, Labib M, Clarke DL, Donkor P, Derbew M, Sani R, Kamara TB, Shrestha S, Nwomeh BC, Wren SM, Price RR, Kushner AL. Surgical care needs of low-resource populations: an estimate of the prevalence of surgically treatable conditions and avoidable deaths in 48 countries. Lancet. 2015 Apr 27;385 Suppl 2:S1. doi: 10.1016/S0140-6736(15)60796-6. Epub 2015 Apr 26. PMID 26313055
- [Background] Lee CHA, Kong JC, Ismail H, Riedel B, Heriot A. Systematic Review and Meta-analysis of Objective Assessment of Physical Fitness in Patients Undergoing Colorectal Cancer Surgery. Dis Colon Rectum. 2018 Mar;61(3):400-409. doi: 10.1097/DCR.0000000000001017. PMID 29377872
- [Background] Lugg ST, Agostini PJ, Tikka T, Kerr A, Adams K, Bishay E, Kalkat MS, Steyn RS, Rajesh PB, Thickett DR, Naidu B. Long-term impact of developing a postoperative pulmonary complication after lung surgery. Thorax. 2016 Feb;71(2):171-6. doi: 10.1136/thoraxjnl-2015-207697. PMID 26769017
- [Background] Hall DE, Arya S, Schmid KK, Carlson MA, Lavedan P, Bailey TL, Purviance G, Bockman T, Lynch TG, Johanning JM. Association of a Frailty Screening Initiative With Postoperative Survival at 30, 180, and 365 Days. JAMA Surg. 2017 Mar 1;152(3):233-240. doi: 10.1001/jamasurg.2016.4219. PMID 27902826
- [Background] Bibo L, Goldblatt J, Merry C. Does preoperative pulmonary rehabilitation/physiotherapy improve patient outcomes following lung resection? Interact Cardiovasc Thorac Surg. 2021 May 27;32(6):933-937. doi: 10.1093/icvts/ivab011. PMID 33907813
- [Background] Bevilacqua Filho CT, Schmidt AP, Felix EA, Bianchi F, Guerra FM, Andrade CF. Risk factors for postoperative pulmonary complications and prolonged hospital stay in pulmonary resection patients: a retrospective study. Braz J Anesthesiol. 2021 Jul-Aug;71(4):333-338. doi: 10.1016/j.bjane.2021.02.003. Epub 2021 Feb 3. PMID 34229858
- [Background] Kutluk AC, Akin H, Ceritoglu A, Kocaturk CI, Bilen S, Sonmezoglu Y, Karapinar K. Is the Outcome of Pulmonary Resections due to Non-Small Cell Lung Cancer in Octogenarian Patients Worse? Ann Thorac Cardiovasc Surg. 2019 Apr 20;25(2):95-101. doi: 10.5761/atcs.oa.18-00206. Epub 2018 Dec 11. PMID 30542000
- [Background] Katsura M, Kuriyama A, Takeshima T, Fukuhara S, Furukawa TA. Preoperative inspiratory muscle training for postoperative pulmonary complications in adults undergoing cardiac and major abdominal surgery. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD010356. doi: 10.1002/14651858.CD010356.pub2. PMID 26436600
- [Background] Westerdahl E, Lindmark B, Eriksson T, Friberg O, Hedenstierna G, Tenling A. Deep-breathing exercises reduce atelectasis and improve pulmonary function after coronary artery bypass surgery. Chest. 2005 Nov;128(5):3482-8. doi: 10.1378/chest.128.5.3482. PMID 16304303
- [Background] Hanada M, Kanetaka K, Hidaka S, Taniguchi K, Oikawa M, Sato S, Eguchi S, Kozu R. Effect of early mobilization on postoperative pulmonary complications in patients undergoing video-assisted thoracoscopic surgery on the esophagus. Esophagus. 2018 Apr;15(2):69-74. doi: 10.1007/s10388-017-0600-x. Epub 2017 Dec 16. PMID 29892929
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Chan SY, Chen CF. Effects of an Active Music Therapy Program on Functional Fitness in Community Older Adults. J Nurs Res. 2020 Oct;28(5):e111. doi: 10.1097/JNR.0000000000000391. PMID 32649395
- [Background] Spagnuolo R, Corea A, Blumetti M, Giovinazzo A, Serafino M, Pagliuso C, Pagnotta R, Curto G, Cosco C, Cosco V, Mancina RM, Garieri P, Papaleo A, Grande L, Barilaro A, Garofalo E, Bruni A, Doldo P. Effects of listening to music in digestive endoscopy: A prospective intervention study led by nursing. J Adv Nurs. 2020 Nov;76(11):2993-3002. doi: 10.1111/jan.14516. Epub 2020 Sep 9. PMID 32901972
- [Background] Ardo NP, Loizzi D, Panariti S, Piccinin I, Sollitto F. Enhanced recovery pathways in thoracic surgery from Italian VATS group: nursing care program. J Thorac Dis. 2018 Mar;10(Suppl 4):S529-S534. doi: 10.21037/jtd.2017.12.85. PMID 29629199
- [Background] Forooghy M, Mottahedian Tabrizi E, Hajizadeh E, Pishgoo B. Effect of Music Therapy on Patients' Anxiety and Hemodynamic Parameters During Coronary Angioplasty: A Randomized Controlled Trial. Nurs Midwifery Stud. 2015 Jun;4(2):e25800. doi: 10.17795/nmsjournal25800. Epub 2015 Jun 27. PMID 26339666
- [Background] Liu Y, Petrini MA. Effects of music therapy on pain, anxiety, and vital signs in patients after thoracic surgery. Complement Ther Med. 2015 Oct;23(5):714-8. doi: 10.1016/j.ctim.2015.08.002. Epub 2015 Aug 4. PMID 26365452
- [Background] Binns-Turner PG, Wilson LL, Pryor ER, Boyd GL, Prickett CA. Perioperative music and its effects on anxiety, hemodynamics, and pain in women undergoing mastectomy. AANA J. 2011 Aug;79(4 Suppl):S21-7. PMID 22403963
- [Background] Calik-Kutukcu E, Saglam M, Vardar-Yagli N, Cakmak A, Inal-Ince D, Bozdemir-Ozel C, Sonbahar-Ulu H, Arikan H, Yalcin E, Karakaya J. Listening to motivational music while walking elicits more positive affective response in patients with cystic fibrosis. Complement Ther Clin Pract. 2016 May;23:52-8. doi: 10.1016/j.ctcp.2016.03.002. Epub 2016 Mar 16. PMID 27157959
- [Background] Kushnir J, Friedman A, Ehrenfeld M, Kushnir T. Coping with preoperative anxiety in cesarean section: physiological, cognitive, and emotional effects of listening to favorite music. Birth. 2012 Jun;39(2):121-7. doi: 10.1111/j.1523-536X.2012.00532.x. Epub 2012 May 17. PMID 23281860
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Zengin S, Kabul S, Al B, Sarcan E, Dogan M, Yildirim C. Effects of music therapy on pain and anxiety in patients undergoing port catheter placement procedure. Complement Ther Med. 2013 Dec;21(6):689-96. doi: 10.1016/j.ctim.2013.08.017. Epub 2013 Sep 1. PMID 24280479
- [Background] Twiss E, Seaver J, McCaffrey R. The effect of music listening on older adults undergoing cardiovascular surgery. Nurs Crit Care. 2006 Sep-Oct;11(5):224-31. doi: 10.1111/j.1478-5153.2006.00174.x. PMID 16983853
- [Background] Ozer N, Karaman Ozlu Z, Arslan S, Gunes N. Effect of music on postoperative pain and physiologic parameters of patients after open heart surgery. Pain Manag Nurs. 2013 Mar;14(1):20-8. doi: 10.1016/j.pmn.2010.05.002. Epub 2010 Dec 22. PMID 23452523
- [Background] Schneider MA. The Effect of Listening to Music on Postoperative Pain in Adult Orthopedic Patients. J Holist Nurs. 2018 Mar;36(1):23-32. doi: 10.1177/0898010116677383. Epub 2016 Nov 10. PMID 29436975
- [Background] Wang Y, Dong Y, Li Y. Perioperative psychological and music interventions in elderly patients undergoing spinal anesthesia: effect on anxiety, heart rate variability, and postoperative pain. Yonsei Med J. 2014 Jul;55(4):1101-5. doi: 10.3349/ymj.2014.55.4.1101. PMID 24954343
- [Background] Ugras GA, Yildirim G, Yuksel S, Ozturkcu Y, Kuzdere M, Oztekin SD. The effect of different types of music on patients' preoperative anxiety: A randomized controlled trial. Complement Ther Clin Pract. 2018 May;31:158-163. doi: 10.1016/j.ctcp.2018.02.012. Epub 2018 Feb 17. PMID 29705448
- [Background] Celebi D, Yilmaz E, Sahin ST, Baydur H. The effect of music therapy during colonoscopy on pain, anxiety and patient comfort: A randomized controlled trial. Complement Ther Clin Pract. 2020 Feb;38:101084. doi: 10.1016/j.ctcp.2019.101084. Epub 2019 Dec 23. PMID 32056820
- [Background] Zhang ZS, Wang XL, Xu CL, Zhang C, Cao Z, Xu WD, Wei RC, Sun YH. Music reduces panic: an initial study of listening to preferred music improves male patient discomfort and anxiety during flexible cystoscopy. J Endourol. 2014 Jun;28(6):739-44. doi: 10.1089/end.2013.0705. Epub 2014 Mar 31. PMID 24548148
- [Background] Canga B, Azoulay R, Raskin J, Loewy J. AIR: Advances in Respiration - Music therapy in the treatment of chronic pulmonary disease. Respir Med. 2015 Dec;109(12):1532-9. doi: 10.1016/j.rmed.2015.10.001. Epub 2015 Oct 19. PMID 26522499
- [Background] Ulubay G, Dilektasli AG, Borekci S, Yildiz O, Kiyan E, Gemicioglu B, Saryal S. Turkish Thoracic Society Consensus Report: Interpretation of Spirometry. Turk Thorac J. 2019 Jan 1;20(1):69-89. doi: 10.5152/TurkThoracJ.2018.180175. PMID 30664428